CLINICAL TRIAL: NCT03788226
Title: A Randomized Phase III Study Comparing POF (Paclitaxel/Oxaliplatin/Leucovorin/5-FU) With SOX/CAPOX/FOLFOX as a Postoperative Adjuvant Chemotherapy for Curatively Resected Stage III Gastric Cancer
Brief Title: A Randomized Phase III Study Comparing POF With SOX/CAPOX/FOLFOX as a Postoperative Adjuvant Chemotherapy for Curatively Resected Stage III Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF 014
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer Stage III
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POF (Experimental): A 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and leucovorin (400 mg/m2), administered simultaneously over a 2-hour infusion period. Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating every 14 days for 12 cycles.
  Interventions: Drug: POF
- CAPOX/SOX/FOLFOX (Active Comparator): CAPOX: IV oxaliplatin given over 120 min at a dose of 130 mg/m2 on day 1, oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days for 8 cycles.
  SOX: Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days for 8 cycles.
  mFOLFOX6: IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-Fluorouracil 400 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 46h every 14 days for 12 cycles.
  Interventions: Drug: CAPOX/SOX/FOLFOX

INTERVENTIONS:
Drug: POF — A 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and leucovorin (400 mg/m2), administered simultaneously over a 2-hour infusion period. Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating every 14 days for 12 cycles.
  Arms: POF
Drug: CAPOX/SOX/FOLFOX — CAPOX: IV oxaliplatin given over 120 min at a dose of 130 mg/m2 on day 1, oral capecitabine 1000 mg/m2 twice daily on days 1 through 14 every 21 days for 8 cycles.
  SOX: Oxaliplatin 130mg/m2 IV on D1 every 21 days and S-1 80mg/m2/day PO [BSA <1.25 40mg bid (total 80mg/day); BSA ≥1.25 - <1.5 50mg bid (total 100mg/day); BSA ≥1.5 60mg bid (total 120mg/day)], divided by two on D1-14 every 21 days for 8 cycles.
  mFOLFOX6: IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-Fluorouracil 400 mg/m2 and IV infusional 5-Fluorouracil 2400 mg/m2 over 46h every 14 days for 12 cycles.
  Arms: CAPOX/SOX/FOLFOX

SUMMARY:
FNF-014 is a randomised, open-label, multicentre, parallel-group, phase 3 study in China to prove superiority of POF over S-1/docetaxel in postoperative adjuvant setting for pStage III gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years.
* Histologically proven in gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction) of stage IIIA, IIIB, IIIC with no evidence of metastatic disease.
* Subjects must be able to take orally.
* R0 resection with D2 lymph-node dissection with al least 15 lymph nodes were examined to ensure adequate disease classification.
* Previously untreated except for the initial gastric resection for the primary lesion.
* ECOG performance status ≦ 1.
* Able to start chemotherapy with 42 days after gastrectomy.
* Hgb ≧ 9 g/dL, WBC 4000-12000/mm3, platelets ≧ 100,000/mm3
* Creatine ≦ upper normal limit (UNL)
* Total bilirubin ≦ 1.5 X UNL
* AST, ALT and ALP ≦ 2.5 x UNL
* Life expectancy estimated than 3 months
* Written informed consent

Exclusion Criteria:

* Active double cancer
* Gastrointestinal bleeding
* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant
* Definite contraindications for the use of corticosteroids
* Any subject judged by the investigator to be unfit for any reason to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | From enrollment to 5 years after treatment
  The time from randomisation to the time of recurrence of the original gastric cancer, development of a new gastric cancer, or death from any cause

SECONDARY OUTCOMES:
overall survival | From enrollment to 5 years after treatment
  The time from the date of randomisation to date of death from any cause
safety (The incidence of chemotherapy related adverse events) | From enrollment to 1 years after treatment
  The incidence of chemotherapy related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Rongbo Lin, Fuzhou, China

IPD SHARING:
Plan to Share IPD: Undecided